CLINICAL TRIAL: NCT04049136
Title: Comparison of Amino-Terminal Pro-Brain Natriuretic Peptide Levels in Healthy Obese and Non-Obese Pregnant Women
Brief Title: NT-proBNP Levels and Obesity in Pregnancy
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: PRO00101213
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2019-08

CONDITIONS: Obesity; Pregnancy Complications; Peripartum Cardiomyopathy
MeSH Terms: conditions — Obesity; Pregnancy Complications; Peripartum Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy pregnant women with BMI <30
  Interventions: Diagnostic Test: NT-proBNP
- Healthy pregnant women with BMI >=30
  Interventions: Diagnostic Test: NT-proBNP

INTERVENTIONS:
Diagnostic Test: NT-proBNP — Measure levels of NT-proBNP in healthy pregnancy women across BMI categories.

SUMMARY:
A screening modality to help categorize obese pregnant women as high or low probability for heart failure would be helpful in the evaluation of the obese pregnant women with dyspnea. Outside of pregnancy, measurement of brain natriuretic peptide (BNP) or amino-terminal pro-brain natriuretic peptide (NT-proBNP) is recommended in the evaluation of acute dyspnea and in the diagnosis of heart failure. During pregnancy, elevated BNP has been associated with adverse cardiovascular events, while normal BNP levels have been observed in healthy pregnancies. While BNP levels outside of pregnancy have been shown to be lower in obese patients variations in BNP levels by body mass index (BMI) in pregnancy have not been studied. Before BNP can be deemed a reliable screening test for heart failure in obese pregnant women, normal BNP values in the setting of obesity and pregnancy need to be established. We therefore propose the following specific aims:

Objective 1: Compare mean plasma NT-proBNP levels in the third trimester, immediately postpartum, and at 4-6 weeks postpartum between obese pregnant women without cardiovascular disease and non-obese pregnant women without cardiovascular disease. We hypothesize that mean plasma NT-proBNP levels in obese pregnant women without pre-existing cardiovascular disease will be significantly lower than levels in non-obese pregnant women.

Objective 2: Assess whether plasma NT-proBNP levels in pregnancy correlate with BMI. We hypothesize that there will be an inverse correlation between plasma NT-proBNP levels and BMI in our pregnant cohort similar to that seen outside of pregnancy.

DETAILED DESCRIPTION:
This study is a prospective, cross-sectional observational study of pregnant women >= 18-years-old receiving prenatal care through the Duke University Health System. Potential study subjects will be approached by obstetric providers or by trained research staff at routine prenatal visits. Approximately 55 subjects will be enrolled, accounting for a potential 10% loss to follow-up.

Women with pre-pregnancy BMI ≥ 30 will be considered obese, while women with BMI <30 will be included in the non-obese control group. Extremely obese (BMI≥40), obese (30≤BMI<40), overweight (25≤BMI<30), and non-obese subjects (BMI<25) will be recruited in a 1:1:1:1 fashion. Subjects will not be matched.

Data collection

Once consent to participate in the study has been obtained and a patient has been deemed eligible to participate, plasma N-terminal pro-brain natriuretic peptide (collected into a PST tube), maternal weight, and systolic and diastolic blood pressure will be collected at the given timepoints:

1. Third-trimester - 27-28 weeks' gestation with third-trimester lab work (CBC, HIV, glucola)
2. Admission to labor and delivery (for labor, rupture of membranes, or scheduled delivery) with admission lab work
3. Immediate postpartum: 24-48 hours postpartum
4. Delayed postpartum (4-6 weeks' postpartum to coincide with postpartum visit)

The following additional data will be collected from the electronic medical record: maternal age, maternal height, maternal pre-pregnancy weight, maternal weight at each time point, best obstetric estimate of due date, patient-reported race/ethnicity, gravida, para, smoking status, mode of delivery, delivery date, date of hospital discharge, minimum and maximum systolic and diastolic blood pressures during labor admission, type of anesthesia used, hemoglobin and hematocrit at 3rd-trimester lab draw, admission, and immediately postpartum (if available), and blood loss at delivery. At each visit, subjects will also be questioned about symptoms and signs of heart failure, including dyspnea on exertion, orthopnea, chest pain, and lower extremity edema.

PST tubes will be collected by trained research staff at the timepoints listed above. These will then be sent to the Duke Clinical Lab for analysis, at which point the samples will be centrifuged and the plasma analyzed for NT-proBNP. NT-proBNP will be analyzed using an electrochemiluminescence immunoassay on the Roche cobas e411 analyzer.

At each study visit time point, subjects will be asked about any symptoms related to heart failire. Should they answer yes to any of the questions, the study team will notify their clinical care team.

ELIGIBILITY:
Eligibility criteria Third-trimester pregnancy (≥27 weeks)

Exclusion criteria Age ≥ 18 years English-speaking Fetal complications

* Fetal anomalies
* Intrauterine fetal demise
* Fetal growth restriction (<5%ile)
* Fetal aneuploidy Maternal complications
* Chronic hypertension (diagnosis pre-dating pregnancy or BP ≥140/90 at <20 weeks gestation)
* Autoimmune disorders (systemic lupus erythematosus, rheumatoid arthritis, Sjogren's)
* Baseline renal disease (baseline Cr >1.0)
* Pre-existing diabetes mellitus
* History of cardiomyopathy or heart failure
* History of cardiac arrest or myocardial infarction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnancy
Study Population: This study is a prospective, cross-sectional observational study of pregnant women >= 18-years-old receiving prenatal care through the Duke University Health System.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
NT-proBNP | 27-29 weeks
  NT-proBNP levels in pregnancy across BMI categories
NT-proBNP | delivery admission
  NT-proBNP levels in pregnancy across BMI categories
NT-proBNP | 24-48 hours postpartum
  NT-proBNP levels in pregnancy across BMI categories
NT-proBNP | 4-6 week postpartum visit
  NT-proBNP levels in pregnancy across BMI categories

CONTACTS AND LOCATIONS:
Overall Officials: Chad A Grotegut, MD, MBA, Principal Investigator — Duke Health
Locations (1):
- Duke Perinatal Durham Clinic, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Denoble AE, Moyett JM, Goldstein SA, Ward CC, Truong T, Erkanli A, James AH, Grotegut CA. Prospective Observational Study of N-terminal Pro-Brain Natriuretic Peptide Levels in Obese and Nonobese Women during Pregnancy. Am J Perinatol. 2023 Apr;40(5):467-474. doi: 10.1055/a-1925-1532. Epub 2022 Aug 16. PMID 35973801